CLINICAL TRIAL: NCT05464589
Title: Effects of Transcutaneous Tibial Nerve Stimulation for Overactive Bladder Symptoms in Adults: A Randomized Control Trial
Brief Title: Effects of Transcutaneous Tibial Nerve Stimulation for Overactive Bladder Symptoms in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Sana Subhan, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SSubhan
Record Dates: First submitted 2022-04-09; First posted 2022-07-19 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Overactive Bladder; Urge Incontinence; Nocturia
Keywords: Lower urinary tract symptoms (LUTS); urge incontinence; overactive detrusor; neuromodulation therapy; nocturia; pelvic floor disease
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge; Nocturia; Lower Urinary Tract Symptoms; Pelvic Floor Disorders

STUDY DESIGN:
Intervention Model Description: It is a randomized control trial. Total 60 patients will be recruited, 30 in each group. Treatment will be allocated using a random number sheet generated by SPSS software version 21. Participants are assigned to one of two groups in parallel for the duration of the study.
Who Masked: Outcomes Assessor
Masking Description: The outcome accessor involved in the clinical trial will be prevented from having knowledge of the interventions to the individual participants of each group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcutaneous Tibial Nerve Stimulation + Pelvic Floor Muscle Strengthening (Experimental): Pelvic floor muscle strengthening through Kegel exercises along with the transcutaneous tibial nerve stimulation.
  Pelvic Floor Muscle-strengthening exercises - Kegels' exercises 15 repetitions, 3 times a day For 6 weeks, daily.
  Transcutaneous Tibial Nerve Stimulation for 30 minutes on the right lower limb 6 sessions, one per week.
  Interventions: Other: Transcutaneous tibial nerve stimulation along with pelvic floor muscle srengthening
- Pelvic Floor Muscle Strengthening (Active Comparator): Pelvic floor muscle strengthening through Kegel exercises.
  Pelvic floor muscle exercises - Kegels; exercises 15 repetitions, 3 times a day For 6 weeks, daily.
  Interventions: Other: Pelvic floor muscles strengthening

INTERVENTIONS:
Other: Transcutaneous tibial nerve stimulation along with pelvic floor muscle srengthening — Pelvic floor muscles strengthening:
  Pelvic floor muscles training involves Kegel's exercises. Kegel exercises improve the function and tone of the pelvic floor. Kegel exercises represent the voluntary contraction and relaxation of the levator ani muscle (principally the pubococcygeus and puborectalis portions), which supports the vagina, bladder, and urethra. The slow contractions help with muscle strengthening.
  Transcutaneous electrical stimulation of Tibial Nerve:
  Transcutaneous Tibial nerve stimulation is a form of treatment technique that involves the use of electrical impulses to address urinary symptoms and target the lower urinary tract.
  Arms: Transcutaneous Tibial Nerve Stimulation + Pelvic Floor Muscle Strengthening
Other: Pelvic floor muscles strengthening — Pelvic floor muscles strengthening:
  Pelvic floor muscles training involves Kegel's exercises. Kegel exercises improve the function and tone of the pelvic floor. Kegel exercises represent the voluntary contraction and relaxation of the levator ani muscle (principally the pubococcygeus and puborectalis portions), which supports the vagina, bladder, and urethra. The slow contractions help with muscle strengthening.
  Arms: Pelvic Floor Muscle Strengthening

SUMMARY:
For overactive bladder symptoms, there are numerous physiotherapy techniques have been found to be beneficial. Transcutaneous electrical stimulation of the tibial nerve is one of those treatment options, that is entirely a non-invasive, easy to apply, and cost-effective technique.

Transcutaneous stimulation of the tibial nerve targets the sacral nerve plexus that contracts the pelvic floor muscles and controls the bladder function.

This research aims to study the effectiveness of transcutaneous tibial nerve stimulation in adults with overactive bladder symptoms along with the conventional physiotherapy for overactive bladder (pelvic floor muscle training through Kegel's exercises) among 60 patients with overactive bladder symptoms on the basis of non-probability purposive sampling technique with screening for study criteria through a consultant urologist. After taking informed consent, all participants will be randomly allocated into two groups. Group A will receive pelvic floor muscles training through Kegels exercises along with transcutaneous electrical stimulation of the tibial nerve and Group B will receive pelvic floor muscles training through Kegels exercises. The treatment duration will of six weeks. Outcomes will be assessed before the start of the treatment and after the end of the treatment sessions.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed overactive bladder
* A total OABSS score of 3 or more and an urgency score of 2 or more
* 30-65 years old

Exclusion Criteria:

* Pregnancy
* Acute urinary tract infection (within 15 days)
* Any surgical procedure for urinary incontinence
* Genito-urinary cancer history
* Stage II pelvic organ prolapse according to pelvic organ prolapse-quantification system
* Lesion on the site of stimulation or around it
* Pelvic pacemakers
* Lower limbs prostheses
* Patients who will not be able to perform Kegel's exercises
* An impaired sensation at the site of stimulation.
* Patients receiving any treatment other than the prescribed medications by the referring physician (that will be the same for all patients of both groups) will be excluded.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
Change in Overactive Bladder Symptom Score from baseline at sixth week | At baseline and after 6 weeks
  OABSS is a validated instrument which evaluates the four cardinal symptoms (day and nighttime frequency, urgency, and urge incontinence) of OAB in a one score. A total OABSS score of 3 or more and an urgency score of 2 or more is the recommended cut-off for diagnosing OAB, and the severity is further divided into mild (total score of 3-5 points), moderate (6-11 points) and severe (12 or more points).
  Patients will be evaluated at baseline and 6 weeks after the intervention through OABSS.

CONTACTS AND LOCATIONS:
Overall Officials: Sana Subhan, DPT, Principal Investigator — Dow University of Health Sciences; Dr. Syed Imran Ahmed, MBBS, FCPS, Study Director — Sindh Institute of Physical Medicine and Rehabilitation; Dr. Muhammad Hammad Mithani, MBBS, FCPS, Study Director — Dow University Hospital; Aftab Ahmed Mirza Baig, DPT, MSAPT, Study Director — Sinsh Institute of Physical Medicine and Rehabilitation
Locations (3):
- Pakistan (3):
  - Dow University Hospital, Karachi, Sindh
  - Dow University of Health Sciences, Karachi, Sindh
  - Sindh Institute of Physical Medicine and Rehabilitation, Karachi, Sindh

REFERENCES:
- [Background] Schreiner L, dos Santos TG, Knorst MR, da Silva Filho IG. Randomized trial of transcutaneous tibial nerve stimulation to treat urge urinary incontinence in older women. Int Urogynecol J. 2010 Sep;21(9):1065-70. doi: 10.1007/s00192-010-1165-6. Epub 2010 May 11. PMID 20458465
- [Background] Lightner DJ, Gomelsky A, Souter L, Vasavada SP. Diagnosis and Treatment of Overactive Bladder (Non-Neurogenic) in Adults: AUA/SUFU Guideline Amendment 2019. J Urol. 2019 Sep;202(3):558-563. doi: 10.1097/JU.0000000000000309. Epub 2019 Aug 8. PMID 31039103
- [Background] Bhide AA, Tailor V, Fernando R, Khullar V, Digesu GA. Posterior tibial nerve stimulation for overactive bladder-techniques and efficacy. Int Urogynecol J. 2020 May;31(5):865-870. doi: 10.1007/s00192-019-04186-3. Epub 2019 Dec 18. PMID 31853597
- [Background] Jacomo RH, Alves AT, Lucio A, Garcia PA, Lorena DCR, de Sousa JB. Transcutaneous tibial nerve stimulation versus parasacral stimulation in the treatment of overactive bladder in elderly people: a triple-blinded randomized controlled trial. Clinics (Sao Paulo). 2020 Jan 10;75:e1477. doi: 10.6061/clinics/2020/e1477. eCollection 2020. PMID 31939564
- [Background] Booth J, Connelly L, Dickson S, Duncan F, Lawrence M. The effectiveness of transcutaneous tibial nerve stimulation (TTNS) for adults with overactive bladder syndrome: A systematic review. Neurourol Urodyn. 2018 Feb;37(2):528-541. doi: 10.1002/nau.23351. Epub 2017 Jul 21. PMID 28731583
- [Background] Ramirez-Garcia I, Blanco-Ratto L, Kauffmann S, Carralero-Martinez A, Sanchez E. Efficacy of transcutaneous stimulation of the posterior tibial nerve compared to percutaneous stimulation in idiopathic overactive bladder syndrome: Randomized control trial. Neurourol Urodyn. 2019 Jan;38(1):261-268. doi: 10.1002/nau.23843. Epub 2018 Oct 12. PMID 30311692
- [Background] Wein AJ, Rovner ES. Definition and epidemiology of overactive bladder. Urology. 2002 Nov;60(5 Suppl 1):7-12; discussion 12. doi: 10.1016/s0090-4295(02)01784-3. PMID 12493342
- [Background] Ouslander JG. Management of overactive bladder. N Engl J Med. 2004 Feb 19;350(8):786-99. doi: 10.1056/NEJMra032662. No abstract available. PMID 14973214
- [Background] Eapen RS, Radomski SB. Review of the epidemiology of overactive bladder. Res Rep Urol. 2016 Jun 6;8:71-6. doi: 10.2147/RRU.S102441. eCollection 2016. PMID 27350947
- [Background] Homma Y, Yoshida M, Seki N, Yokoyama O, Kakizaki H, Gotoh M, Yamanishi T, Yamaguchi O, Takeda M, Nishizawa O. Symptom assessment tool for overactive bladder syndrome--overactive bladder symptom score. Urology. 2006 Aug;68(2):318-23. doi: 10.1016/j.urology.2006.02.042. PMID 16904444